CLINICAL TRIAL: NCT06169709
Title: Diagnosis and Experiences From Women With ADHD; an International Survey
Brief Title: An Online Survey for Women With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: Parnassia Groep (Other)
Responsible Party: Principal Investigator, Danielle de Graaf, Principal investigator, Parnassia Groep
Other Study IDs: Survey Female ADHD
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this exploratory study following a cross-sectional online survey in women with ADHD is to

1. describe overall experiences regarding ADHD symptoms, diagnosis, treatment, sources of support, and any perceived barriers on those domains;
2. determine which life domains are most affected by ADHD symptoms;
3. calculate the prevalence of reported health conditions within the following domains: circulatory system, endocrine or metabolic system, gastrointestinal system, genitourinary system, musculoskeletal system, nervous system, respiratory system, skin, reproductive system, cancer, psychiatric conditions, COVID-19, sensory sensitivity, menstrual cycle, and sleep;
4. identify topics that women with ADHD would like to see studied in future research.

DETAILED DESCRIPTION:
Rationale: In clinical practice, the investigators see that ADHD affects women differently than men. It has become clear that a better understanding of ADHD in girls and women is needed to improve their longer-term wellbeing and functional and clinical outcomes.

Objective: The primary endpoint is to describe the overall experience of women with ADHD regarding ADHD symptoms, diagnosis, treatment, and any perceived barriers relating to these domains. The investigators also want to determine the effects of ADHD symptoms on day-to-day life across various life domains. Moreover, the investigators want to determine the prevalence of reported health conditions.

Study design: This is an exploratory study following a cross-sectional online survey.

Study population: Women (aged >18 years) with ADHD.

Intervention (if applicable): Not applicable.

Main study parameters/endpoints: In women with ADHD, the investigators want to 1) describe overall experiences regarding ADHD symptoms, diagnosis, treatment, sources of support, and any perceived barriers on those domains; 2) determine which life domains are most affected by ADHD symptoms; 3) calculate the prevalence of reported health conditions within the following domains: circulatory system, endocrine or metabolic system, gastrointestinal system, genitourinary system, musculoskeletal system, nervous system, respiratory system, skin, reproductive system, cancer, psychiatric conditions, COVID-19, sensory sensitivity, menstrual cycle, and sleep; 4) identify topics that women with ADHD would like to see studied in future research.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This survey is the first to study experiences and health of women with ADHD internationally, and results will provide insights and leads for all involved with diagnosis and treatment of these women. Risks of participation are considered low. Participants might consider certain questions triggering, but are always free to skip questions and stop the survey.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a woman
* Aged 18 or above
* Have ADHD (both diagnosed by a health professional and self-diagnosed)

Exclusion Criteria:

* People who are not able to read, understand, or sign the information letter or informed consent form are excluded from participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who identify as women.
Study Population: The survey is aimed at women (or people who identify as women) over 18 years with ADHD (both self-diagnosed and diagnosed by a health professional).
Sampling Method: Non-Probability Sample
Enrollment: 5893 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
To describe the overall experiences, thoughts, and perspectives of women with ADHD, including domains of ADHD diagnosis and symptoms, ADHD and other health conditions, menstrual cycle, conflict tactics and romantic relationships, and sleep. | 50 minutes
  A self-developed questionnaire. The sections on demographic information, ADHD diagnosis, ADHD diagnosis & symptoms and menstrual cycles are constructed for the purpose of this survey. Moreover, the questionnaire contains sections from the Ultrashort screener for adult ADHD, the Holland Sleep Disorder Questionnaire and the Conflict Tactics scale 2.

SECONDARY OUTCOMES:
To identify topics for further research and ways of improving healthcare (e.g. the diagnostic process or effective treatment) for women with ADHD | 50 minutes
  Questions are included in the questionnaire described for outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Kooij, Prof. dr., Principal Investigator — PsyQ
Locations (1):
- Parnassia Groep, The Hague, Netherlands

IPD SHARING:
Plan to Share IPD: No